CLINICAL TRIAL: NCT00146484
Title: A Randomized Controlled Trial of Two Versus Three Daily Insulin Injections in Children and Adolescents With New Onset Type 1 Diabetes Mellitus
Brief Title: A Study of Two Versus Three Daily Injections in Children and Adolescents With Newly Diagnosed Type 1 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Hospital of Eastern Ontario (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHEO RI cc9993
Record Dates: First submitted 2005-09-06; First posted 2005-09-07 (Estimated); Last update posted 2005-09-07 (Estimated); Status verified 2005-09

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Diabetes Mellitus, Type 1; Child; Adolescent; Disease Management; Newly Diagnosed; Hemoglobin A, Glycosylated
MeSH Terms: conditions — Diabetes Mellitus, Type 1

INTERVENTIONS:
Drug: Twice Daily versus Three Times Daily Insulin Injections

SUMMARY:
The optimal insulin regimen for children and adolescents with newly diagnosed type 1 diabetes remains unknown. The purpose of this study is to determine whether a split evening injection regimen (insulin injections before breakfast, supper and bedtime) leads to better glucose control and quality of life than twice daily insulin in children and adolescents with new onset diabetes.

DETAILED DESCRIPTION:
The optimal insulin regimen for children and adolescents with newly diagnosed type 1 diabetes remains unknown. No published studies have examined the effectiveness of a split evening (three times daily) injection regimen in this group of patients. Indeed, because the first few years of diabetes management are the easiest (due to a "honeymoon" period characterised by residual insulin secretion), the potential for any benefit from more intensive management (i.e., three daily injections) may be small during this period. In addition, the intensity of the initial insulin regimen may be an important determinant of quality of life, family functioning, and subsequent compliance with diabetes regimens. A randomized controlled trial has been designed to test the hypothesis that a split evening injection regimen leads to better glycemic control and quality of life than twice daily insulin in children and adolescents with new onset diabetes.

ELIGIBILITY:
Inclusion Criteria:

* New onset type 1 diabetes
* Less than 48 hours since first insulin injection
* Child and/or parent able to read and write English
* Family intends to continue treatment at our institution for the next two years
* Informed consent from adolescents greater than 16 years of age, or if less than 16 years, informed consent from the parent/guardian with assent from the child.

Exclusion Criteria:

* Chronic medical conditions other than treated hypothyroidism or mild asthma
* Concerns of the diabetes team regarding future treatment adherence making twice daily insulin preferable to the split evening injection regimen (e.g., cognitive impairment, severe family dysfunction).

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100
Dates: Start 1996-04; Study Completion 2001-01

PRIMARY OUTCOMES:
* Hemoglobin A1c over the first 24 months of diabetes

SECONDARY OUTCOMES:
* Frequency of hypoglycemia (mild and severe) over the first 24 months of diabetes
* Frequency of morning hyperglycemia over the first 24 months of diabetes
* Residual c-peptide at two years post diagnosis (stimulated c-peptide post Sustacal challenge)
* Diabetes Quality of Life (DQOLY) over the first 24 months of diabetes
* Family Functioning (Family Environment Scale)over the first 24 months of diabetes

CONTACTS AND LOCATIONS:
Overall Officials: Margaret L Lawson, MD, Principal Investigator — Children's Hospital of Eastern Ontario
Locations (1):
- Children's Hospital of Eastern Ontario, Ottawa, Ontario, Canada